CLINICAL TRIAL: NCT04904055
Title: Value-based Formulary-Essentials: Testing and Expanding on Value in Prescription Drug Benefit Design
Brief Title: Evaluating the Impact of a Value-based Prescription Drug Formulary
Acronym: VBF-e
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Donaghue Medical Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 218066
Record Dates: First submitted 2021-05-17; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Value-Based Health Insurance
Keywords: Cost Sharing / economics; Formularies as Topic; Insurance, Health / economics; Value-Based Health Insurance / economics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Value-based Formulary Beneficiaries: enrolled in the value-based formulary
  Interventions: Other: Value-based Formulary
- Standard Formulary Beneficiaries: enrolled in a standard (i.e., non-value-based formulary)

INTERVENTIONS:
Other: Value-based Formulary — Prescription drug formulary tiers informed by estimated value
  Groups: Value-based Formulary Beneficiaries

SUMMARY:
The objective of this study is to evaluate the impact of the value-based formulary on patient out-of-pocket spending and health plan spending as well as the impact of the value-based formulary on medication use, emergency department visits, hospitalizations, and outpatient office visits.

ELIGIBILITY:
Inclusion Criteria:

* Individuals:

  * aged 0-64
  * Continuously enrolled in an employer-sponsored health plan for at least 12 months (with one-month allowable gap) prior to the index date

    * For individuals in the exposed group, the index date is defined as the start date of value-based formulary implementation at the employer group level
    * For individuals in the control group, the index date is defined as the index date of the matched exposed individual
* Employer groups:

  * that transition to the value-based formulary if they transitioned all enrollees in that employer group (no individual selection)

Exclusion Criteria:

- Individuals with:

* missing gender information
* missing zip code level demographics at all member months

Ages: 0 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All individuals who satisfy the eligibility criteria are included.
Sampling Method: Non-Probability Sample
Enrollment: 36333 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Total spending for prescription drugs | From 24 months before insurance transition until up to 36 months after transition
  Impact of value-based formulary on patient out-of-pocket plus health plan spending on prescription drugs per member per month

SECONDARY OUTCOMES:
Patient out-of-pocket spending for prescription drugs | From 24 months before insurance transition until up to 36 months after transition
  Impact of value-based formulary on patient out-of-pocket spending for prescription drugs per member per month
Health plan spending for prescription drugs | From 24 months before insurance transition until up to 36 months after transition
  Impact of value-based formulary on health plan spending for prescription drugs per member per month
Total healthcare spending | From 24 months before insurance transition until up to 36 months after transition
  Impact of value-based formulary on total healthcare spending per member per month
Number of emergency department visits | From 24 months before insurance transition until up to 36 months after transition
  Impact of value-based formulary on number of emergency department visits per member per month
Number of days in hospital | From 24 months before insurance transition until up to 36 months after transition
  Impact of value-based formulary on number of days in hospital per member per month
Number of outpatient office visits | From 24 months before insurance transition until up to 36 months after transition
  Impact of value-based formulary on number of outpatient office visits per member per month
Days supply of medication | From 24 months before insurance transition until up to 36 months after transition
  Impact of value-based formulary on days supply of medication per member per month

CONTACTS AND LOCATIONS:
Overall Officials: Kai Yeung, PharmD, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available per data use agreement.

REFERENCES:
- [Derived] Yeung K, Cruz M, Tsiao E, Watkins JB, Sullivan SD. Drug use and spending under a formulary informed by cost-effectiveness. J Manag Care Spec Pharm. 2023 Nov;29(11):1175-1183. doi: 10.18553/jmcp.2023.29.11.1175. PMID 37889867

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT04904055/SAP_000.pdf